CLINICAL TRIAL: NCT06092307
Title: SARcopenia in Patients With ChrOnic PANcreatitis: the SARCOPAN Study
Acronym: SARCOPAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5507
Record Dates: First submitted 2023-09-20; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Electric Impedance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic pancreatitis (Experimental): adult patients aged 18-65 years with a diagnosis of chronic pancreatitis
  Interventions: Diagnostic Test: Bioelectrical impedance; Diagnostic Test: Handgrip strength test; Diagnostic Test: muscle ultrasound.

INTERVENTIONS:
Diagnostic Test: Bioelectrical impedance — Resistance, reactance, phase angle,free-fat mass, body cell mass, body cell mass index and total body will be recorded
Diagnostic Test: Handgrip strength test — Handgrip strength test using a hydraulic hand dynamometer and sit-to-stand test will be performed.
Diagnostic Test: muscle ultrasound. — The following ultrasound parameters will be evaluated: radial, ulnar, rectus femoris, rectus abdominis and medial gastrocnemius muscle thickness and echo intensity with gray-scale-index; rectus femoris muscle cross sectional area; gastrocnemius muscle fiber length and pennation angle.

SUMMARY:
Sarcopenia is a complex multifactorial syndrome which could be present in older age (primary sarcopenia) or earlier in chronic disease (secondary sarcopenia). Evidence of the prevalence and incidence of sarcopenia in chronic pancreatitis is lacking, as well as studies which correlate sarcopenia to evolution of chronic pancreatitis.The main aim of this study is to evaluate whole body composition, sarcopenia, dynamic force tests, laboratory data at different stages of chronic pancreatitis. The accuracy of bioimpedance analysis and muscle ultrasound in the diagnosis of sarcopenia will also be assessed.

DETAILED DESCRIPTION:
INTRODUCTION Sarcopenia is a complex multifactorial syndrome which could be present in older age (primary sarcopenia) or earlier in chronic disease (secondary sarcopenia). It is associated with worse prognosis in terms of quality of life, morbidity, and mortality. Among causes of secondary sarcopenia, chronic inflammation, endocrine dysregulation, malnutrition, and malabsorption are some of the most important factors. All these conditions are present in chronic pancreatitis (CP) with or without endocrine or exocrine pancreatic insufficiency (EPI). Chronic pancreatitis is characterized by chronic inflammation of the gland, with acinar and ductal destruction and progressive replacement of injured pancreatic tissue by fibrotic tissue. As a result, pancreatic functions gradually decline and exocrine pancreatic insufficiency and pancreatogenic diabetes emerge. Evidence of the prevalence and incidence of sarcopenia in chronic pancreatitis is lacking, as well as studies which correlate sarcopenia to evolution of chronic pancreatitis. In a recent metanalysis, Kuan et la reported a prevalence of sarcopenia in CP ranging from 17 to 62%. Assessing sarcopenia and body composition in patients with chronic pancreatitis is an important prognostic factors as its impact on clinical outcome.The gold standard to diagnose sarcopenia is the measurement of muscle mass using computed tomography or magnetic resonance. Primary limitations of these procedures are the radiation exposure and costs, respectively. Muscle ultrasonography may be the ideal method for evaluating both muscle quality and quantity since it is inexpensive, easy to replicate, and unobtrusive. Different studies demonstrated a significant correlation between muscle ultrasound and muscle mass assessed with gold standard technique. To investigators' knowledge, no study has analysed the application of ultrasonography in the assessment of sarcopenia in chronic pancreatitis.

The main aim of this study is to evaluate whole body composition, sarcopenia, dynamic force tests, laboratory data at different stages of chronic pancreatitis. The accuracy of bioimpedance analysis and muscle ultrasound in the diagnosis of sarcopenia will also be assessed.

Materials and methods Ninety-eight patients with diagnosis of chronic pancreatitis will be enrolled in this prospective study. Inclusion criteria are age between 18 and 65 years, and CT, or MRI into precedent maximum 12 months. Exclusion criteria include age less than 18 or older than 65 and lack of informed consent.

Based on CT and MRI, CP will be classified according to Cambridge classification. Diagnosis of EPI will be defined according to fecal elastase <200 mg/g .

Serum nutritional markers associated with CP and PEI amylase, lipase, vitamin D, vitamin B12, folate, total protein, albumin, total cholesterol, HDL cholesterol, triglycerides will be recorded.

Concerning body composition, weigh, height, and BMI will be recorded. Bioelectrical impedance will be performed, and following parameters will be recorded: resistance, reactance, phase angle, free-fat mass, body cell mass, body cell mass index and total body.

Cross-sectional skeletal muscle Area (SMA), visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT) and intramuscular adipose tissue (IMAT) will be evaluated on a transversal scan at the level of third lumbar vertebra (L3). SMI will be calculated as SMA/height ratio. Sex relating SMI cut off offs will be used to established sarcopenia diagnosis (male <56.44 cm2/m2, female <46.56 cm2/m2).

Handgrip strength test using a hydraulic hand dynamometer and sit-to-stand test will be performed to assess dynamic muscle force.

All patients will undergo a muscle ultrasound. The following ultrasound parameters will be evaluated: radial, ulnar, rectus femoris, rectus abdominis and medial gastrocnemius muscle thickness and echo intensity with gray-scale-index; rectus femoris muscle cross sectional area; gastrocnemius muscle fiber length and pennation angle.

Statistical analysis This is monocenter, prospective, non-pharmacological trial. Nominal or ordinal variables will be presented as frequencies and percentages. Mean, standard deviation, median and 95% confidence intervals will be calculated for continuous variables. Comparison between means/median will be investigated with Mann-Whitney test or t-Student test. Association between sarcopenia and demographic and disease characteristic will be assessed using Chi-square and Fisher exact test.

Furthermore, multivariate analysis will be performed. Correlation will be established using Pearson or Spearman correlation coefficient. The area under the receiver operating characteristic (AUROC) will be calculated to evaluate performance of muscle ultrasound and bioelectrical impedance and specific cut off will be determined calculating the Youden index. A p value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* diagnosis of chronic pancreatitis
* age between 18 and 65 years,
* abdominal CT or MRI into precedent maximum12 months.

Exclusion Criteria:

* age less than 18 or older than 65 years
* lack of informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
sarcopenia prevalence in chronic pancreatitis | three months
  skeletal muscle index (SMI) = skeletal muscle Area (SMA)/height
whole body composition in chronic pancreatitis | three months
  measurement of skeletal muscle mass through bioelectrical impedance
dynamic muscle force | three months
  Handgrip strength test using a hydraulic hand dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy